CLINICAL TRIAL: NCT05458284
Title: Acupuncture for Taxane-Induced Peripheral Neuropathy Prevention (ATP): A Phase II Randomized, Placebo Controlled Trial
Brief Title: The Effect of Acupuncture on Nerve Pain Caused by Taxane (Chemotherapy) Treatment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-197
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Taxane-Induced Peripheral Neuropathy
Keywords: Acupuncture; Peripheral Neuropathy; 22-197
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real acupuncture (RA) (Active Comparator): Real Acupuncture weekly till taxane completion
  Interventions: Procedure: Real Acupuncture
- sham acupuncture (SA) (Placebo Comparator): Sham Acupuncture weekly till taxane completion
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Procedure: Real Acupuncture — Real Acupuncture weekly till taxane completion
  Arms: real acupuncture (RA)
Other: Sham Acupuncture — Sham Acupuncture weekly till taxane completion
  Arms: sham acupuncture (SA)

SUMMARY:
Some people experience a side effect while they are receiving taxane called taxane-induced peripheral neuropathy (TIPN). TIPN is pain in the arms and legs due to nerve damage caused by cancer treatment and may interfere with quality of life. The purpose of this study is to learn if acupuncture can prevent TIPN from getting worse. Acupuncture is a medical technique that involves insertion of very thin needles into specific areas on the body. We will compare real acupuncture (RA) to placebo (sham) acupuncture (SA). SA is done like RA, but will use different needles and target different sites or places on the body than RA. We are comparing RA to SA to learn whether RA can prevent TIPN from getting worse while receiving taxane.

DETAILED DESCRIPTION:
The study will include two phases. The first phase is the screening phase, in which patients with early stage breast cancer undergoing taxane therapy will consent and receive TIPN screening each week till they develop grade 1 or higher by CTCAE criteria. The patients with TIPN grade 1 or higher will then be consented to the intervention phase, in which patients will be randomized to receive either weekly real or sham acupuncture treatment using a standardized, semi-fixed protocol developed in our preliminary studies to improve TIPN pain. The participant may also participate in Part 2 of the study if they begin to experience TIPN but do not participate in Part 1.

ELIGIBILITY:
Inclusion Criteria:

Screening Phase:

* English or Spanish-proficient men and women aged ≥18 years
* Histological diagnoses of invasive carcinoma of the breast
* Plan to receive curative intent chemotherapy regimen containing 12 weeks weekly paclitaxel or nab-paclitaxel as standard of care

Intervention Phase:

* TIPN grade ≥1 based on the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, developed while receiving taxane
* ≥ 4 4 weeks of either weekly paclitaxel or nab-paclitaxel, or paclitaxel or abraxane with dosing every 2-3 weeks planned, as standard of care and at treating physician's discretion
* Willing to adhere to requirement that no new pain medication or dose changes be taken throughout the first 12 weeks of the study period
* Willing to adhere to all study-related procedures, including randomization to one of the two possible acupuncture treatments

Exclusion Criteria:

Screening Phase:

* Pre-existing peripheral neuropathy within 28 days of screening consent
* Currently taking anti-neuropathy medication such as gabapentin, pregabalin, duloxetine or glutamine

Intervention Phase:

* Currently taking anti-neuropathy medication such as gabapentin, pregabalin, duloxetine or glutamine
* Use of acupuncture for symptom management within 28 days of intervention consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 80 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Scale (NPS) | at 4 weeks
  Evaluate the effectiveness of real acupuncture versus sham acupuncture in preventing TIPN progression as measured by the Neuropathic Pain Scale (NPS) in patients with early stage breast cancer who are receiving curative intent weekly taxane containing regimen and who have grade ≥ 1 TIPN

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm